CLINICAL TRIAL: NCT05521191
Title: A Phase 1b, Double-Blind, Placebo-Controlled, Multiple Ascending Dose and an Open-Label Fixed-Dose Study in Patients With Autosomal Dominant Polycystic Kidney Disease to Evaluate the Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of RGLS8429
Brief Title: A Study of RGLS8429 in Patients With Autosomal Dominant Polycystic Kidney Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regulus Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: RGLS8429-02
Record Dates: First submitted 2022-08-24; First posted 2022-08-30 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease; ADPKD; Polycystic Kidney, Autosomal Dominant
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Intervention Model Description: The study will consist of two parts. Part A will consist of three sequential cohorts of approximately 12 subjects each randomized centrally to receive RGLS8429 or placebo by subcutaneous injection every other week (Q2W) x 7 doses (approximately 36 subjects total). Part B will be an open-label fixed dose cohort of up to 30 subjects. .
Who Masked: Participant, Investigator
Masking Description: This study will have two parts. Part A is the double-blind, randomized, placebo-controlled study. Part B is the open-label fixed-dose study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- RGLS8429 (Experimental): The randomized,double blind part of the study (Part A) will consist of three sequential cohorts of approximately 12 subjects each randomized centrally to receive RGLS8429 or placebo by subcutaneous injection every other week (Q2W) x 7 doses (36 subjects total).
  * Cohort 1: first dose level of RGLS8429 or placebo
  * Cohort 2: second dose level of RGLS8429 or placebo
  * Cohort 3: third dose level of RGLS8429 or placebo
  Interventions: Drug: RGLS8429
- Placebo (Experimental): The randomized double blind part of the study (Part A) will consist of three sequential cohorts of approximately 12 subjects each randomized centrally to receive RGLS8429 or placebo by subcutaneous injection every other week (Q2W) x 7 doses (36 subjects total).
  * Cohort 1: first dose level of RGLS8429 or placebo
  * Cohort 2: second dose level of RGLS8429 or placebo
  * Cohort 3: third dose level of RGLS8429 or placebo
  Interventions: Drug: Placebo
- Open Label Fixed Dose RGLS8429 (Experimental): The open-label fixed dose part of the study (Part B and Cohort 4) will consist of a single cohort of up to 30 subjects each receiving 300 mg RGLS8429.
  Interventions: Drug: RGLS8429

INTERVENTIONS:
Drug: RGLS8429 — Solution for subcutaneous injection
  Arms: Open Label Fixed Dose RGLS8429; RGLS8429
Drug: Placebo — Solution for subcutaneous injection
  Arms: Placebo

SUMMARY:
Primary Objectives

* To assess the safety and tolerability of RGLS8429
* To assess the impact of RGLS8429 on ADPKD biomarkers

Secondary Objectives

* To assess the impact of RGLS8429 on height-adjusted total kidney volume (htTKV)
* To characterize the pharmacokinetic (PK) properties of RGLS8429
* To assess the impact of RGLS8429 on renal function

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled multiple ascending dose and an open-label fixed-dose Phase 1b study consisting of two parts, Part A and Part B. In Part A, multiple ascending doses of RGLS8429 or placebo will be administered via subcutaneous injection to subjects with ADPKD to evaluate the safety, tolerability, pharmacodynamics and pharmacokinetics of RGLS8429. In Part B, a fixed-dose of RGLS8429 will be administered via subcutaneous injection to subjects with ADPKD to evaluate the safety, tolerability, pharmacodynamics and pharmacokinetics of RGLS8429.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female ADPKD patients, 18 to 70 years old
2. Class 1C, 1D, or 1E Mayo Imaging Classification of ADPKD (based upon either the MRI obtained during screening, or a prior MRI obtained within 5 years of screening with documented Mayo classification)
3. eGFR between 30 to 90 mL/min/1.73 m2
4. Body mass index (BMI) 18 to 35 kg/m2
5. Must understand and consent to the study procedures explained in the ICF and be willing and able to comply with the protocol

Key Exclusion Criteria:

1. Administration of tolvaptan in the 28 days before randomization
2. Subject is mentally incapacitated or has significant emotional problems
3. Any medical condition or social circumstance that, in the opinion of the Investigator, may make the subject unlikely to complete the study or comply with study procedures and requirements; or may pose a risk to the subject's safety
4. History or presence of alcoholism or drug abuse within the past 2 years prior to screening
5. Only one kidney or kidney transplant recipient
6. Participation in another clinical trial and/or exposure to any investigational drug or approved therapy for investigational use within 28 days or 5 half-lives of the investigational drug's dosing, whichever is longer, prior to dosing. The 28-day or 5-half-life windows will be calculated from the date of the last dosing in the previous study to Day 1 of the current study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of RGLS4829: Incidence of AEs | Baseline to Day 113
  Incidence of adverse events over time
Impact of RGLS8429 on ADPKD biomarkers | Baseline to Day 113
  Change from baseline in PC1, PC2, NGAL, and KIM-1 urine biomarkers

SECONDARY OUTCOMES:
Impact of RGLS8429 on height-adjusted total kidney volume (htTKV) | Baseline to Day 113
  Change from baseline in htTKV
Pharmacokinetic properties of RGLS8429: Cmax | Baseline to Day 113
  Maximum observed concentration (Cmax) of RGLS8429
Pharmacokinetic properties of RGLS8429: Tmax | Baseline to Day 113
  Time to maximum observed concentration (Tmax) of RGLS8429
Pharmacokinetic properties of RGLS8429: t½ | Baseline to Day 113
  Half-life of RGLS8429 (t½)

CONTACTS AND LOCATIONS:
Overall Officials: Rekha Garg, MD, Study Director — Regulus Therapeutics
Locations (21):
- United States (21):
  - Centricity Research Phoenix Multispecialty, Mesa, Arizona
  - Academic Medical Research Institute, Los Angeles, California
  - Yale Nephrology Outpatient Clinic, New Haven, Connecticut
  - Mayo Clinic - Florida, Jacksonville, Florida
  - Elixia, Orlando, Florida
  - Southeastern Clinical Research Institute, LLC, Augusta, Georgia
  - CARE Institute, Boise, Idaho
  - CARE Institute, Chubbuck, Idaho
  - The Idaho Kidney Institute, Idaho Falls, Idaho
  - University of Chicago, Chicago, Illinois
  - Research by Design, LLC, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center Jared Grantham Kidney Institute, Kansas City, Kansas
  - Witchita Nephrology Group, PA, Wichita, Kansas
  - University of Maryland School of Medicine, Nephrology, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - St. Clair Nephrology Research, Roseville, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Northeast Clinical Research Center, Bethlehem, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Swedish Center for Comprehensive Care, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] Tekendo-Ngongang C, Gleeson JG, Mignon L. Treating the Untreatable: Antisense Oligonucleotides as an Individualized Therapy for Rare Genetic Kidney Diseases. J Am Soc Nephrol. 2024 Dec 1;35(12):1774-1777. doi: 10.1681/ASN.0000000532. Epub 2024 Sep 27. No abstract available. PMID 39331470